CLINICAL TRIAL: NCT02930213
Title: The Core Body Temperature Rhythms:A Promising Indicator of Distinguishing MCS From UWS
Brief Title: The Core Body Temperature Rhythms: Distinguishing MCS From UWS
Status: Completed | Type: Observational
Sponsor: Jing Wang (Other)
Responsible Party: Sponsor-Investigator, Jing Wang, Principal Investigator, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Other Study IDs: CX2014128
Record Dates: First submitted 2016-09-29; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Disorders of Consciousness
Keywords: unresponsive wakefulness syndrome; minimally conscious state; circadian rhythms; free-running period
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, the core body temperature of 7 disorders of consciousness ( DOC ) patients were measured every 2 hour for 168 h .

DETAILED DESCRIPTION:
Living beings have multicomponent biological rhythms. There was a research recorded 24-h virations in electroencephalographic patterns. In normal subjects, the circadian rhythms of core body temperature is close to 24 h. When the interference of environmental and mental elements were eliminated, circadian rhythm shows the endogenous circadian rhythm of body acquiescently (>24h ), which is also called free-running period.

Measuring the continuous external auditory canal temperature of 4 unresponsive wakefulness syndrome (UWS) and 3 minimally conscious state(MCS) on the fluorescent lamp surrounding every 2 hours for 168 hours starting at 00:00 on the first day to address circadian capabilities.

Researchers expected to see the difference between MCS and UWS.

ELIGIBILITY:
Inclusion Criteria:

* patients in minimally conscious state
* patients with stable condition
* patients free of sedative drugs and Na+ or Ca++ blockers (e.g., carbamazepine) or NMDA receptor antagonist (e.g., dextromethorphan)

Exclusion Criteria:

* premorbid neurology antecedent
* patients in coma or vegetative state
* patients < 1 months after the acute brain injury

Ages: 39 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators chossen patients with UWS or MCS.The subjects include 4 UWS and 3 MCS.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measuring the continuous external auditory canal temperature | Continuous temperature measurements for 168 hours (8days)
  VS patients have core body temperature periods which are longer than 24 hours; whereas MCS patients are shorter than 24 hours.